CLINICAL TRIAL: NCT05640466
Title: Reduction and Fixation of Metatarsal Neck Fracture by Metaizeau's Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hussien Sedik Mohamed, Orthopedic Surgery Resident, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohagu1
Record Dates: First submitted 2022-11-22; First posted 2022-12-07 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Displaced Metatarsal Neck Fracture

STUDY DESIGN:
Masking Description: Single intervention no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patient with displaced metatarsal head fractures (Other): A Kirschner wire with its distal end is placed showing a small bend into the medullar cavity through the lateral margin of the proximal metaphysis of the affected metatarsal using a 5mm skin incision at that level. The skin incision was made over the interosseus space, so as to use one incision for the two neighbouring metatarsal bones. The diameter of the Kirschner wires to be used should be related to the size of the fractured metatarsal medullar cavity. Kirschner wire will be driven anterograde, with the help of an X-ray image intensifier.
  Subsequently, the wire will be rotated 180 to direct its end to the dorsum of the foot so as to provoke a translation effect on the metatarsal head in order to obtain the head reduction, and maintained this reduction with the Kirschner wire.
  Interventions: Device: Reduction and fixation of metatarsal neck fracture by metaizeau's technique

INTERVENTIONS:
Device: Reduction and fixation of metatarsal neck fracture by metaizeau's technique — Reduction and fixation of metatarsal neck fracture by metaizeau's technique

SUMMARY:
Metatarsal fractures represent 3-7% of all fractures of the body and 35% of fractures of the foot and have a rate of 75 new cases per 10,000 persons per year.

The goal of treatment is to achieve a correct reduction of fracture, to avoid prolonged disability and preservation of both soft tissues and bony alignment.

Metaizeau's technique in these fracture of the metatarsal bone respects the soft tissues surrounding the fracture and the periosteum at the fracture site.

DETAILED DESCRIPTION:
Metatarsal fractures represent 3-7% of all fractures of the body and 35% of fractures of the foot and have a rate of 75 new cases per 10,000 persons per year.

Metatarsal fractures have been considered of little importance by many authors over the years, and have received little attention. That is why little literature about operative management of metatarsal fractures can be found (apart from the first and fifth metatarsal bones).

Generally, these are non-displaced fractures. When these fractures show some displacement, reasonable alignment must be obtained because the metatarsals' capability for remodelling is extensive but not infinite.

Displaced metatarsal neck fractures are usually treated by means of retrograde Kirschner wires, which generally requires an open reduction at the fracture site due to the difficulty of reducing the metatarsal head.

Metaizeau's technique can be applied to reduce the displaced metatarsal head distally from the fracture in an easier way and to keep the fracture site closed, as compared with retrograde Kirschner wires method . Open reduction was unnecessary in all cases. This technique permitted correct control of the distal fracture fragment, obtained good reduction of the metatarsal heads without opening the fracture site, and with no lesion of the capsuloligamentous complex of metatarsophalangeal joint. Metaizeau's technique is a valid alternative to retrograde method.

The goal of treatment is to achieve a correct reduction of fracture, to avoid prolonged disability and preservation of both soft tissues and bony alignment. Metaizeau's technique in these fracture of the metatarsal bone respects the soft tissues surrounding the fracture and the periosteum at the fracture site.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with displaced fracture neck of the 2nd, 3rd or 4th metatarsal

Exclusion Criteria:

* Poly_traumatized patient .
* Patient with fracture first and fifth metatarsal bone .
* Fracture shaft metatarsal bone , first MB, fifth MB.
* Open fractures of the foot .
* Intraarticular fracture of metatarsals .
* Lisfranc fracture .
* Segmental fracture of the metatarsals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Central metatarsal fractures: a review and current concepts — https://www.mattioli1885journals.com/index.php/actabiomedica/article/view/9724
- See also: Management of Talar Body Fractures — https://link.springer.com/article/10.4103/ortho.IJOrtho_563_17
- See also: AOFAS Functional Scoring After Antegrade K Wires Fixation of Multiple Metatarsal Neck Fracture: A Case Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8822033/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants came to sohag university hospital
Pre-assignment Details: no participant excluded
Groups:
- Adult Patient With Displaced Metatarsal Head Fractures: A Kirschner wire with its distal end is placed showing a small bend into the medullar cavity through the lateral margin of the proximal metaphysis of the affected metatarsal using a 5mm skin incision at that level. The skin incision was made over the interosseus space, so as to use one incision for the two neighbouring metatarsal bones. The diameter of the Kirschner wires to be used should be related to the size of the fractured metatarsal medullar cavity. Kirschner wire will be driven anterograde, with the help of an X-ray image intensifier.
  Subsequently, the wire will be rotated 180 to direct its end to the dorsum of the foot so as to provoke a translation effect on the metatarsal head in order to obtain the head reduction, and maintained this reduction with the Kirschner wire.
  Reduction and fixation of metatarsal neck fracture by metaizeau's technique: Reduction and fixation of metatarsal neck fracture by metaizeau's technique
Period: Overall Study
Arm/Group | Adult Patient With Displaced Metatarsal Head Fractures
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Patient With Displaced Metatarsal Head Fractures
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 20
  Unknown or Not Reported | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 20

OUTCOME MEASURES:

1. Primary Outcome: Time of Union
Description: Time taken from operation till full fracture union
Time Frame: 8 weeks postoperatively
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Adult Patient With Displaced Metatarsal Head Fractures
Number analyzed (Participants) | 20
weeks | 5.8 (1.48)

2. Primary Outcome: Time to Range of Motion (ROM) Start
Description: Time taken from operation till starting range of motion (ROM)
Time Frame: 8 weeks post-operatively
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Adult Patient With Displaced Metatarsal Head Fractures
Number analyzed (Participants) | 20
weeks | 3.5 (0.51)

ADVERSE EVENTS:
Time Frame: 4 months postoperative
Arm/Group | Adult Patient With Displaced Metatarsal Head Fractures
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patient With Displaced Metatarsal Head Fractures (N=20)
stifness foot (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patient With Displaced Metatarsal Head Fractures (N=20)
Bone infection (Musculoskeletal and connective tissue disorders) | 0 (0)

LIMITATIONS AND CAVEATS:
The small number sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT05640466/Prot_SAP_000.pdf